CLINICAL TRIAL: NCT04395937
Title: Effects of Submaximal Regular Physical Exercise on Quality of Life, Symptomatic Control, and Bronchial and Systemic Inflammatory Markers in Patients With Persistent Asthma
Brief Title: Effects of Regular Submaximal Exercise on Asthma Control and Quality of Life in Patients With Persistent Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Renaud Louis, Professor Doctor, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B707202042981
Record Dates: First submitted 2020-05-04; First posted 2020-05-20 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2021-11

CONDITIONS: Chronic Asthma
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- respiratory physiotherapy (Active Comparator): exercises to improve the way of breathing
  Interventions: Other: exercises
- respiratory physiotherapy and physical exercises (Experimental): intensity determined by the VO2max measured during ergospirometric measure
  Interventions: Other: exercises
- control group (No Intervention)

INTERVENTIONS:
Other: exercises — One hour twice a week to practice respiratory exercises, postural exercises, muscular exercises
  Arms: respiratory physiotherapy; respiratory physiotherapy and physical exercises

SUMMARY:
The effects of regular exercise on asthma control has not yet been well demonstrated.

The aim of this study is to investigate the impact of submaximal physical exercise on quality of life, on symptomatic control, and on bronchial and systemic inflammatory markers in patients with persistant asthma.

DETAILED DESCRIPTION:
While it is well known that intense physical exercise can generate bronchospasm and limit exercise performance, it recently appeared that regular physical exercise practiced aerobically could improve the clinical status of asthmatic patients.

The investigators are planning a 12-week randomized controlled study to assess the effect of regular aerobic exercise on quality of life, asthma control, bronchial hyperresponsiveness and bronchial and systemic inflammation in patients with persistent asthma

The hypothesis is that regular physical exercise increases control and quality of life and reduces inflammation and bronchial hyperresponsiveness compared to simple physiotherapy sessions.

ELIGIBILITY:
Inclusion Criteria:

* asthmatic patient
* aged 18- 90 years
* ACQ > 1.5
* stable background treatment comprising at least one inhaled corticosteroid or an anti-leukotriene

Exclusion Criteria:

* IMC > 35
* severe osteoarthritis of the knees and hips
* unstable angor
* Severe uncontrolled hypertension

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Asthma Quality of Life Questionnaire (AQLQ) | 3 months
  A disease-specific health-related quality of life instrument that taps both physical and emotional impact of disease 32 items with 2-week recall, 4 different domains : Symptoms (11 items), Activity Limitation (12 items, 5 of which are individualized), Emotional Function (5 items), and Environmental Exposure (4 items) 7-point Likert scale (7 = not impaired at all - 1 = severely impaired) Scores range 1-7, with higher scores indicating better quality of life. Change from Baseline AQLQ at 3 months
Asthma Control Questionnaire (ACQ) | 3 months
  A simple questionnaire to measure the adequacy of asthma control and change in asthma control which occurs either spontaneously or as a result of treatment.
  7 items; 1 week recall (for items on symptoms and rescue inhaler use) ACQ has a multidimensional construct assessing symptoms (5 items--self-administered) and rescue bronchodilator use (1 item-self-administered), and FEV1% (1 item) completed by clinic staff 7-point scale (0=no impairment, 6= maximum impairment for symptoms and rescue use; and 7 categories for FEV1%) Scores range between 0 (totally controlled) and 6 (severely uncontrolled). Change from Baseline ACQ at 3 months
FEV1 (Forced Expiratory volume in 1 second) | 3 months
  Change from Baseline FEV1 at 3 months
fall in FEV1 during ergospirometric measurement | 3 months
  Change from Baseline fall in FEV1 during ergospirometric measurement
Amount of eosinophils and neutrophils in sputum | 3 months
  Change from baseline in amount of eosinophils and neutrophils in sputum
FeNo (fractional exhaled nitric oxide) | 3 months
  change from baseline FENO at 3 months
PC20M (measures the concentration of metacholine necessary to bring down the FEV1 by 20% compared to its base value) | 3 months
  Change from baseline PC20M at 3 months
Vo2max (maximum oxygen consumption) | 3 months
  change from baseline Vo2Max at 3 months
PMA (Maximum aerobic power) | 3 months
  change from baseline PMA at 3 months
sputum cell counts | 3 months
  change from baseline
Hospital Anxiety and depression scale (HAD) | 3 months
  The questionnaire comprises seven questions for anxiety and seven questions for depression For each item, 4 response modes coded from 0 to 3. The anxiety and depression items are alternating. In addition, an alteration in the order of the ratings was carried out to avoid biases linked to their repetition.
  An overall score is calculated by adding the 14 items but also 2 subtotals corresponding to the 2 subscales. The higher the scores, the higher the symptomatology.
  From 0 to 7 : absence of anxiety disorders and depressive disorders From 8 to 10 : anxiety and depressive disorders suspected From 11 to 21 : severe anxiety and depressive disorders
Asthma control test (ACT) | 3 months
  change from baseline A questionnaire to determine if patient's asthma symptoms are well controlled. A score varying between 1 and 5 is assigned to each question. A score varying between 1 and 5 is assigned to each question. The higher the total score, the better the asthma is controlled From 1 to 14 : Uncontrolled asthma From 15 to 19 : Partially Controlled Asthma From 20 to 25 : Well controlled asthma
FVC (Forced Vital Capacity) | 3 months
  FVC is the greatest total amount of air the patient can forcefully breathe out after breathing in as deeply as possible Change from Baseline FVC1 at 3 months
TLC (Total Lung Capacity) | 3 months
  It is the total volume of air in the lungs after a maximal inspiration change from baseline TLC at 3 months
DLCO (Diffusing Capacity of the Lung for Carbon Monoxide) | 3 months
  Measures the efficiency of the gas transfer characteristics of the lungs change from baseline DLCO at 3 months
KCO (transfer coefficient of the lung for carbon monoxide) | 3 months
  change from baseline KCO at 3 months
FRC (Functional Residual Capacity) | 3 months
  The volume of air present in the lungs at the end of passive expiration Change from baseline FRC at 3 months
RV (Residual Volume) | 3 months
  It is the amount of air remaining in the lungs after a maximal expiration Change from baseline RV at 3 months
sGaw (Specific airway conductance) | 3 months
  Change from baseline sGaw at 3 months
maximal inspiratory power | 3 months
  Measured in KPa Change from baseline
maximal expiratory power | 3 months
  Measured in KPa Change from baseline
isometric force of long finger grasp | 3 months
  measured using a Jamar dynamometer change from baseline
maximum isometric force of the quadriceps | 3 months
  measured using a dynamometer Change from baseline
VOCs | 3 months
  volatils organics compounds change form baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Liege, Liège, Liege, Belgium